CLINICAL TRIAL: NCT06883201
Title: Application of Patient Blood Management in the Oncology Patient Affected by Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Campus Bio-Medico University (Other); Umberto I Hospital, Frosinone Italy (Other)
Responsible Party: Sponsor
Other Study IDs: RS1796/22
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with breast cancer who have received neoadjuvant chemotherapy or not: Perform a preoperative evaluation through laboratory screening (complete blood count with reticulocyte count, iron balance, vitamin B12 and folate) and prescribe, in case of documented deficiency anemia, a therapy with hematinics. The therapy of choice in most cases of iron deficiency is parenteral ferric carboxymaltose

SUMMARY:
Evaluation of the percentage of transfusions in patients with breast cancer undergoing surgery after preventive treatment with haematinics.

DETAILED DESCRIPTION:
Preoperative anemia treatment is fundamental in Patient Blood Management (PBM) programs, a multidisciplinary and multimodal strategy that improves clinical outcomes based on the patient's blood resource, promoting strategies to optimize hematopoiesis in candidates for elective surgery, in order to significantly reduce the use of blood products, addressing all modifiable transfusion risk factors before it is even necessary to consider the use of transfusion therapy itself. Treatment with intravenous iron reduces the transfusion risk and consequently the adverse events related to the transfusion itself.

Nothing is specified in this regard for cancer patients; very often these patients come to surgery presenting an anaemic state that often requires correction with red blood cell transfusion. The aim of this clinical study is to prevent the number of perioperative transfusions in patients with breast cancer who have undergone or not undergone neoadjuvant chemotherapy and with Hb values lower than or equal to 11 g/dl, who are candidates for destructive and/or reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* patients diagnosed with histologically confirmed breast cancer and whether or not they have undergone neoadjuvant chemotherapy;
* patients who are candidates for destructive and reconstructive breast surgery or not;
* Hb values less than or equal to 11 g/dL and/or transferrin saturation less than or equal to 20%;
* written informed consent.

Exclusion Criteria:

* patients with known allergies to ferric carboxymaltose or its excipients;
* ferritin values greater than 500 ng/ml;
* patients unable to sign consent and comply with procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who have undergone or not undergone neoadjuvant chemotherapy and with Hb values lower than or equal to 11 g/dl, candidates for destructive and/or reconstructive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of transfusions | 18 months
  To evaluate the percentage, in number of transfusions in patients affected by breast cancer, candidates for destructive and/or reconstructive breast surgery after preventive treatment with haematinics

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy